CLINICAL TRIAL: NCT05690100
Title: Clinical Evaluation of the Use of Ozone Gel Versus Hyaluronic Acid Gel on Palatal Wound After Free Gingival Graft Harvesting: A Randomized Controlled Clinical Trial
Brief Title: Evaluation of the Use of Ozone Gel Versus Hyaluronic Acid Gel on Palatal Wound Healing .
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hisham Tarek Mahmoud Ahmed, The Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OZVHA
Record Dates: First submitted 2022-12-26; First posted 2023-01-19 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Palate; Wound
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ozone Gel (Experimental): Ozone is a potent oxidant with marked antimicrobial activity and the potential to act as a metabolic and host immune modulator.The routes of ozone administration are topical and regional for both gaseous and aqueous forms .Ozone gel is contains ozonated extra virgin olive oil and Arnica montana extract, containing essential fatty acids Ozone gel was claimed to have analgesic (Tasxdemir et al,2016) and anti-inflammatory effect its high content of essential fatty acids and the effect of ozone, natural extra virgin olive oil (I. Lezcano,et al.2000). Ozone gel has a beneficial role in wound healing, Its wound healing properties may be due to enhancing blood circulation and immune response.(M.colombo et,al 2019), Generic name : GeliO3 Dosage form : Gel Frequency/Duration : Once on this interval : 0,3,7,14
  Interventions: Drug: GeliO3
- Hyaluronic Acid 0.2% (Experimental): HA was Known for hygroscopicity that allows it to maintain conformational stiffness and to retain water.(Yıldırım et al., 2017b) .Another major feature is viscoelasticity that provides stability and elasticity to tissues and delays penetration of viruses and bacteria (Finn, Schow and Schneiderman, 1992) .
  In periodontology, HA has been advocated as monotherapy(Hammad et al., 2011) or as an adjunct to non-surgical and/or surgical (Fawzy El-Sayed et al., 2012) periodontal treatment to reduce inflammation and promote wound healing.
  HA gel was used in two different concentrations 0.2% and 0.8% versus negative control in the management of post-operative pain after FGG surgery and it was found effective with more superior results for the 0.2% concentration (Yıldırım et al., 2017b).
  Generic name : GingiGel Dosage form : Gel Frequency/Duration : Once on this interval : 0,3,7,14
  Interventions: Drug: Gingi gel

INTERVENTIONS:
Drug: GeliO3 — Anti-inflammatory Gel which has a beneficial role on wound healing
  Arms: Ozone Gel
Drug: Gingi gel — Anti-inflammatory Gel which has a beneficial role on wound healing
  Arms: Hyaluronic Acid 0.2%

SUMMARY:
To compare the effect of Ozone Gel versus Hyaluronic acid gel 0.2% applied to palatal donor site in post-operative pain reduction after free gingival graft harvesting.

DETAILED DESCRIPTION:
To compare the effect of Ozone Gel versus Hyaluronic acid gel 0.2% applied to palatal donor site in post-operative pain reduction , Color match , Wound size closure after free gingival graft harvesting.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mucogingival defects scheduled for free gingival graft
* Systemically healthy

Exclusion Criteria:

* Smokers
* Occlusal trauma at site of graft
* Pregnancy and lactation
* Patients allergic to the used agents
* Severe gagging reflex

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Post Operative Pain | 14 days
  Post operative pain measured directly through VAS score with 0 means no pain and 10 means the maximum pain or indirectly by analgesics consumption by the patient

SECONDARY OUTCOMES:
Color Match | 42 days
  the color of the palatal mucosa will be assessed by comparing it with that of the adjacent and opposite side by using the objective VAS (VAS score 0-10) represented by a continuous line, by a clinician blinded to the treatment group assignment.
  A score of 0 indicates no color match, and a score of 10 indicates excellent color match with the adjacent tissues.
Wound Size | 42 days
  Wound size decrease/closure

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M barbari, Study Director — Cairo University; Dalia M Ghalwash, Study Chair — Cairo University; Nesma M Shemais, Study Chair — Cairo University; Hisham Ahmed, Principal Investigator — Cairo University

REFERENCES:
- [Background] Yildirim S, Ozener HO, Dogan B, Kuru B. Effect of topically applied hyaluronic acid on pain and palatal epithelial wound healing: An examiner-masked, randomized, controlled clinical trial. J Periodontol. 2018 Jan;89(1):36-45. doi: 10.1902/jop.2017.170105. PMID 28914592